CLINICAL TRIAL: NCT06702917
Title: Wide Coverage GSI Cardiac Data Collection
Brief Title: GSI Cardiac on Revolution Apex - US
Status: Recruiting | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: SA-000042
Record Dates: First submitted 2024-11-22; First posted 2024-11-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Coronary Computed Tomographic Angiography; Myocardial Infarction (MI); Cardiac Catheterization
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Cohort A: Undergoing a standard of care CCTA
  Interventions: Device: GSI Cardiac Scan; Other: Standard of Care CCTA
- Cohort B: Known history of heart attack (myocardial infarction) or undergoing a standard of care cardiac catheterization due to known disease
  Interventions: Device: GSI Cardiac Scan; Other: Research CCTA

INTERVENTIONS:
Device: GSI Cardiac Scan — The investigational GSI Cardiac scan will take place immediately ("back-to-back acquisition") following the single energy, non-GSI CCTA. The GSI Cardiac scan takes around 1 minute.
  A subset of Cohort B's participants who are eligible due to a history of heart attack will have the investigational GSI Cardiac scan 10-15 minutes after the end of the CCTA scan.
Other: Standard of Care CCTA — The standard of care scan will be a single-energy, non-GSI CCTA. Any pre-contrast screening (such as kidney function or pregnancy testing) will follow the site's standard operating procedures. The administration of contrast media (either IV or oral) and any cardiac medications used to control heart rate will be prescribed per the site's standard operating procedures. All contrast and cardiac medications will be FDA approved and used in accordance with its approval.
  Groups: Cohort A
Other: Research CCTA — The research scan will be a single-energy, non-GSI CCTA. Any pre-contrast screening (such as kidney function or pregnancy testing) will follow the site's standard operating procedures. The administration of contrast media (either IV or oral) and any cardiac medications used to control heart rate will be prescribed per the site's standard operating procedures. All contrast and cardiac medications will be FDA approved and used in accordance with its approval.
  Groups: Cohort B

SUMMARY:
The goal of this clinical data collection study is to collect raw CT scan data using a new GSI Cardiac mode on GE HealthCare's Revolution Apex CT system.

Two groups of participants will be enrolled:

A) Participants scheduled to undergo a Coronary CT Angiography (CCTA) as part of their standard of care

B) Participants scheduled to undergo a cardiac catheterization or have a history of heart attack

Participants in Group A will:

-Have a standard of care CCTA immediately followed by a research GSI Cardiac scan

Participants in Group B will:

-Have a research CCTA immediately followed by a research GSI Cardiac scan

Both groups will be in the study for approximately 1 day. There are no follow-up visits after the day of scan.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in this study if they meet the following criteria:

1. Who are ≥18 years of age;
2. Able to sign and date the informed consent form; AND,
3. Cohort A: Undergoing a scheduled clinically indicated CCTA; OR,
4. Cohort B: Known history of myocardial infarction or undergoing a clinically indicated cardiac catheterization due to known pathology.

Exclusion Criteria:

Subjects may be excluded from participating in study if they meet any of the following criteria:

1. Who are pregnant or lactating;
2. Who were previously enrolled in this study;
3. Anyone with known or suspected allergy to iodinated contrast agents;
4. Anyone with known or suspected renal insufficiency as determined by site medical personnel;
5. Who are in need of urgent or emergent care;
6. Who have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the subject;
7. Who are unwilling to have GEHC personnel present for the CT exam; AND,
8. Cohort A: Undergoing a scheduled clinically indicated CCTA for anatomy assessment (aberrant origin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of adults that are 18-years of age or older, and who are undergoing either a scheduled CCTA, a scheduled cardiac catheterization due to known history of pathology or is a patient with known history of myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluable GSI Cardiac Raw Scans | 12 months
  Number of participants whose GSI Cardiac scan is deemed evaluable (i.e., no issues with participant motion or contrast administration and/or timing).

SECONDARY OUTCOMES:
Safety Assessment | 12 months
  Number of Adverse Events and/or Serious Adverse Events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Thomsen, Study Director — GE Healthcare
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No